CLINICAL TRIAL: NCT07326033
Title: Efficacy and Safety of Allogenic Cultured Adipose-derived Mesenchymal Stromal Cell Injections on MoUth Fibrosis and Handicap in Patients With Systemic sclEroderma
Acronym: A-MUSE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC31/22/0258; 2024-518516-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-04; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Systemic Scleroderma
Keywords: Systemic Scleroderma; microstomia; oral health-related quality of life; oral pathology; regenerative medicine; allogenic cultured adipose-derived stromal cells
MeSH Terms: conditions — Scleroderma, Systemic; Microstomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AdMSC (Experimental): Patients will be standard of care (physiotherapy and daily self-administered exercises) and receive allogeneic AdMSC injection in the perioral (lips) region.
  Interventions: Drug: AdMSC
- Placebo (Placebo Comparator): Patients will be standard of care (physiotherapy and daily self-administered exercises) and receive placebo injections in the perioral (lips) region
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AdMSC — At day 0, patients will have AdMSC injections in perioral region. Patients will be followed-up for 24 weeks
  Arms: AdMSC
Drug: Placebo — At day 0, patients will have placebo injections in perioral region. Patients will be followed-up for 24 weeks
  Arms: Placebo

SUMMARY:
Orofacial manifestations and microstomia are a frequent complication in systemic sclerosis (SSc) with a major impact on oral hygiene, dental care and quality of life. Peri-oral injection of allogeneic cultured adipose-derived stromal cells constitutes a promising approach to treat scleroderma-induced mouth fibrosis where no alternative therapy is validated. The aim of this phase 2 study is to compare efficacy and safety of perioral injection of allogeneic cultured adipose-derived stromal cells (AdMSC) versus placebo to improve oro-facial fibrosis in patients with systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥18 years of age,
* Patient with systemic scleroderma according to the 2013 ACR/EULAR classification criteria,
* Mouth Handicap in Systemic Sclerosis Scale (MHISS) score more than or equal to 20 (0-48),
* Rodnan skin score on the face more than or equal to 1,
* Maximal mouth opening of less than 40 mm (distance between the dental arches)
* Patient must have provided written informed consent prior to enrolment,
* Patient must be able to understand their requirements of participating in the protocol.
* Patient affiliated to a social security system.

Exclusion Criteria:

* Patient participating in a clinical trial or having participated in a clinical trial within the previous 3 months,
* Injection of botulinum toxin within 4 weeks prior to "inclusion visit",
* Patient who underwent autologous hematopoietic stem cell transplantation (HSCT) within less than 1 year,
* Local active labial herpes virus within 1 week prior to "inclusion visit",
* Patients with an indication for intensification by autologous HSCT (according to EBMT guidelines and national MATHEC-SFGMTC guidelines),
* History of cancer in the last five years, except for successfully excised basal cell/squamous cell carcinoma, or successfully excised early melanoma of the skin. Subjects, who had a successful tumor resection or radiation or chemotherapy more than 5 years prior to inclusion and no recurrence, may be enrolled in the study,
* Radio- or chemotherapy in progress,
* Females who are pregnant or breastfeeding or plan to be or do so during the course of this study,
* Women of childbearing potential (WOCBP) who are sexually active and unwilling to use an adequate birth control method,
* Vulnerable patient (persons deprived of their liberty by judicial or administrative decision, persons undergoing psychiatric treatment, persons admitted to a health or social establishment for purposes other than research) according to article L1121-6 of the Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Mouth Handicap in Systemic Sclerosis scale (MHISS) | Day 0, 12 weeks after injection
  the change in the Mouth Handicap in Systemic Sclerosis scale (MHISS) between baseline and week 12. An improvement of at least 5 points will be considered clinically significant

SECONDARY OUTCOMES:
Safety of treatment | Day 0, 4, 12 and 24 weeks after injection
  The safety throughout the course of the study (until week 24 since baseline) will be assessed by monitoring adverse events, serious adverse events and injection site reactions.
Efficacy on oral function by facial scanners | Day 0, 4, 12 and 24 weeks after injection
  Efficacy on oral function is a composite measure derived from the change in maximum interincisal distance and mouth perimeter by facial scanners with digital acquisition of the patient's face in just a few seconds
Efficacy on orofacial handicap | Day 0, 4, 12 and 24 weeks after injection
  Efficacy on orofacial handicap is a composite measure derived from change in Opening, Dryness and Aesthetic the 3 subscales of the MHISS
Patient satisfaction | Day 0, 4, 12 and 24 weeks after injection
  the patients will be asked to fill in a simple questionnaire where their degree of satisfaction could be expressed by a composite measure derived by a semiquantitative score (unsatisfied, mildly/moderately satisfied, rather satisfied, and very satisfied), Scleroderma Health Assessment Questionnaire (sHAQ), Oral Health Assessment Tool (OHAT), Burden of Face Affected questionnaire (BOFA) and EQ-5D-5L
Oral habits and hygiene | Day 0 and 24 weeks after injection
  Change in oral habits and hygiene is a composite measure derived from oral health and hygiene questionnaire
oral microbiota | Day 0, 12 and 24 weeks after injection
  Change in oral microbiota mesuared in unstimulated saliva
Plaque index | Day 0, 12 and 24 weeks after injection
  Change in Plaque index (reflecting the ability to maintain oral hygiene)
Change in decayed missing filled teeth | Day 0 and 24 weeks after injection
  Change in decayed missing filled teeth (DMFT) index : a commonly used index validated by the WHO to assess oral status and the examinator simply counts the number of decayed, missing (due to caries or periodontal disease) and restored/filled teeth.
Change in mandibular tracking | Day 0, 4, 12 and 24 weeks after injection
  Change Mandibular tracking is a composite measure derived from mandibular tracking and articular and neuro-muscular activity. Mandibular tracking and neuro-muscular activity will be measured with electrodes positioned in order to assess muscular activity at rest, muscle activity during mouth closure as well as during extreme movement of mouth opening and closing, mandibular propulsion and deduction. Muscle contraction synchronism and contraction efficacy will also be measured as well as the 3-dimensional innoclusion space and mandibular movement during swallowing
Posture by stabilometry | Day 0, 12 and 24 weeks after injection
  Change posture by stabilometry
psycho-social aspects and oro-facial pains | Day 0, 4, 12 and 24 weeks after injection
  Change in psycho-social aspects and oro-facial pains is a composite measure derived from EDAS21, Epworth and Combadazou-Destruhaut questionnaire
Rodnan skin score | Day 0, 12 and 24 weekds after injection
  Change in modified Rodnan skin score
Dry mouth syndrome | Day 0, 4, 12 and 24 weeks after injection
  Change in dry mouth syndrome is a composite measure derived from the change in Xerostomia Inventory questionnaire , in salivary flow, in the salivary pH and Salivary pH
Efficacy on aesthetics | Day 0, 4 , 12 and 24 weeks after injection
  the efficacy on aesthetics assessed by Standardized two-dimensional photographs or face scan
Immunomonitoring of vascular and antifibrotic biomarkers | Day 0 and 12 weekds after injection
  Immunomonitoring of vascular and antifibrotic biomarkers (V5. Endothelin-1, Endostatin, Endogline, Angiotensin I and II, Tie 1 and 2, VEGF, sICAM-1, sVCAM, E-selectin, CXCL4) measured in blood samples

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Bordeaux Hospital, Bordeaux
  - Dijon Hospital, Dijon
  - Montpellier Hospital, Montpellier
  - Nantes Hospital, Nantes
  - Toulouse Hospital, Toulouse